CLINICAL TRIAL: NCT05545618
Title: Biological Interconnection of Brain Neurobiological Activity With Atherosclerotic Plaque Vulnerability and the Prognostic Value
Brief Title: Brain-heart Interaction in Coronary Plaque Stability and Cardiovascular Events
Acronym: Blueprint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2022-9-15
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA imaging with 18F-FDG-PET/CT assessment: Group of patients with 18F-FDG-PET/CT imaging and Coronary Computed Tomographic Angiography within 90 days
  Interventions: Diagnostic Test: CCTA and 18F-FDG-PET/CT

INTERVENTIONS:
Diagnostic Test: CCTA and 18F-FDG-PET/CT — 18F-FDG-PET/CT imaging and comprehensive assessment of coronary plaque with CCTA within 90 days

SUMMARY:
The effect of brain-heart interaction remains unclear. The study aims to investigate the biological interconnection between brain neural activity and coronary plaque morphological and inflammatory features, as well as their connection with clinical outcomes.

DETAILED DESCRIPTION:
Brain neural activity assessed by resting amygdalar activity (AmygA) can predict cardiovascular events. However, its biological interconnection with plaque vulnerability i is not fully understood. Coronary computed tomographic angiography (CCTA) is a non-invasive technique that enables comprehensive assessment of morphological characteristics of coronary atheroma and estimates the level of plaque instability. Recently, perivascular fat attenuation index (FAI) enables assessment of coronary inflammation by analyzing changes of perivascular adipose tissue attenuation in CCTA.

18F-fluorodeoxyglucose-positron emission tomography/computed tomography (18F-FDG-PET/CT) enables simultaneous estimation of multi-system activities including brain neural activity and hematopoiesis.

The present study aims to use ¹⁸F-FDG PET/CT to assess the AmygA, and to investigate its association with CCTA assessed plaque morphological and inflammatory features as well as their ability in predicting future cardiovascular disease events.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: greater than 20
* 2) Patients either absence of prior cancer or remission from cancer for at least 1 year prior to imaging and throughout the follow-up period;
* 3) Patients absence of acute or chronic inﬂammatory or autoimmune disease at the time of imaging;
* 4) Patients with CCTA performed within 90 days of 18F-FDG PET/CT scan as part of routine clinical practice
* 5) Patients with diameter stenosis >30% by CCTA but without coronary revascularization

Exclusion Criteria:

* 1) Complex coronary lesion (ostial lesion, unprotected left main lesion, chronic total occlusion, grafted vessels, etc)
* 2) Coronary lesion with heavy calcification
* 3) Chronic renal insufficiency (Serum creatinine >2.0mg/dL)
* 4) Severe liver dysfunction (aspartate transaminase or alanine transferase > 5 times of upper normal limit)
* 5) Pregnancy or potential pregnancy
* 6) Life expectancy less than 5 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent clinically indicated 18F-FDG PET/CT and with CCTA performed within 90 days of 18F-FDG PET/CT scan will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation Between amygdalar activity (neurobiological activity) and bone marrow hematopoiesis (hematopoietic activity) | at the index imaging
  Amygdalar target-to-background ratio (TBR) = Amygdalar standardized uptake value (SUV) / Temporal lobe SUV Bone marrow TBR = Bone marrow SUV / Jugular vein SUV Correlation between amygdalar activity (neurobiological activity) and bone marrow hematopoiesis (hematopoietic activity) will be assessed
Correlation Between amygdalar activity (neurobiological activity) and high-risk plaque | at the index imaging
  High-risk plaque features will be assessed by CCTA including positive remodeling (PR, defined as lesion diameter/reference diameter ≥1.1), low attenuation plaque (LAP, defined as a focal central area of plaque with an attenuation density of <30 Hounsfield Units), spotty calcification (SC, defined as focal calcification within the coronary artery wall <3mm in maximum diameter), and the "napkin ring" sign (defined as a central area of low attenuation plaque that had a peripheral rim of high attenuation).
  Correlation Between amygdalar activity and number of high-risk plaque features will be assessed.
Correlation Between amygdalar activity (neurobiological activity) and coronary inflammation | at the index imaging
  Coronary inflammation will be assessed by FAI. Correlation Between amygdalar activity and FAI will be assessed
Major adverse cardiac events | 5 years after index imaging
  Death from coronary heart disease, nonfatal myocardial infarction or hospitalization for unstable angina.

SECONDARY OUTCOMES:
Cardiovascular death, or nonfatal myocardial infarction | 5 years after index imaging
  Cardiovascular death, or nonfatal myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University
Locations (4):
- China (4):
  - Fuwai Hospital, Beijing
  - Shanghai Zhongshan Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Universal Medical Imaging Diagnostic, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tawakol A, Ishai A, Takx RA, Figueroa AL, Ali A, Kaiser Y, Truong QA, Solomon CJ, Calcagno C, Mani V, Tang CY, Mulder WJ, Murrough JW, Hoffmann U, Nahrendorf M, Shin LM, Fayad ZA, Pitman RK. Relation between resting amygdalar activity and cardiovascular events: a longitudinal and cohort study. Lancet. 2017 Feb 25;389(10071):834-845. doi: 10.1016/S0140-6736(16)31714-7. Epub 2017 Jan 12. PMID 28088338
- [Background] Tawakol A, Osborne MT, Wang Y, Hammed B, Tung B, Patrich T, Oberfeld B, Ishai A, Shin LM, Nahrendorf M, Warner ET, Wasfy J, Fayad ZA, Koenen K, Ridker PM, Pitman RK, Armstrong KA. Stress-Associated Neurobiological Pathway Linking Socioeconomic Disparities to Cardiovascular Disease. J Am Coll Cardiol. 2019 Jul 2;73(25):3243-3255. doi: 10.1016/j.jacc.2019.04.042. PMID 31248544
- [Derived] Dai N, Tang X, Weng X, Cai H, Zhuang J, Yang G, Zhou F, Wu P, Liu B, Duan S, Yu Y, Guo W, Ju Z, Zhang L, Wang Z, Wang Y, Lu B, Shi H, Qian J, Ge J. Sex Differences in Coronary Inflammation and Atherosclerosis Phenotypes in Response to Imaging Marker of Stress-Related Neural Activity. Circ Cardiovasc Imaging. 2024 Feb;17(2):e016057. doi: 10.1161/CIRCIMAGING.123.016057. Epub 2024 Feb 20. PMID 38377235